CLINICAL TRIAL: NCT01594086
Title: Effects of Green Tea Consumption on Homocysteine Metabolism and Cognitive Dysfunction in Elderly: An Exploratory Clinical Study
Brief Title: Effects of Green Tea Consumption on Homocysteine Metabolism and Cognitive Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Shizuoka (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT201201; 24220501 (Other: Ministry of Health, Labor and Welfare)
Record Dates: First submitted 2012-05-01; First posted 2012-05-08 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Cognitive Impairment
Keywords: green tea; aging; atherosclerosis; homocysteine; cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- green tea powder (Experimental): Natural green tea powder
  Interventions: Dietary Supplement: green tea powder

INTERVENTIONS:
Dietary Supplement: green tea powder — Consuming 2 g/day of green tea powder in three times divided for 3 months

SUMMARY:
Green tea contains catechins and theanine as major ingredients and has been reported to have various beneficial influences on human health. It is reported that the drinking green tea is inversely associated with serum homocysteine level in elderly. However the effect of green tea consumption on cognitive dysfunction is not clinically clarified. The purpose of this study is to investigate the effects of green tea consumption on homocysteine metabolism and cognitive dysfunction in elderly with impaired cognitive function.

DETAILED DESCRIPTION:
Elderly people with impaired cognitive function go on increasing year by year with the coming aged society. Among them, the Alzheimer disease is a major cause of the illness, which is progressively worse, has no fundamental curable therapy, and induces the burdens of caregivers as well as the health insurance and national budget. Recently, homocysteine metabolism is reported to be related to atherosclerosis in aging, and draw attention as the etiology of cognitive dysfunction in elderly.

Green tea contains catechins and theanine as main ingredients. These components are reported to have anti-atherogenic action and effect on improving cognitive dysfunction. However, clinical evidence for homocysteine metabolism and cognitive dysfunction has not been clarified. Therefore, in this study, the investigators attempted to investigate the effects of green tea consumption on homocysteine metabolism and cognitive dysfunction in elderly with impaired cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Obtained written informed consent before participation
* Possible to consume green tea powder
* Possessing cognitive dysfunction; MMSE score less than 30
* Possible not to take any supplement possessing anti-oxidizing effect; i.e., vitamin A, C, E, β-carotene

Exclusion Criteria:

* Possessing allergy to green tea
* Possessing severe cardiac, respiratory, renal, or hepatic dysfunction
* Possessing severe anemia
* Diagnosed as inadequate to participate in the study by doctor

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Changes in the serum homocysteine levels | between baseline and 3 months after
  Changes in the serum homocysteine levels before and after the intervention

SECONDARY OUTCOMES:
Changes in serum lipid levels | between baseline and 3 months after
  Changes in serum lipid levels before and after the intervention
Changes in serum folic acid levels | between baseline and 3 months after
  Changes in serum folic acid levels before and after the intervention
Changes in mini mental state examination (MMSE) scores | between baseline and 3 months after
  Changes in mini mental state examination (MMSE) scores before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yamada, Hiroshi, Study Chair — University of Shizuoka
Locations (1):
- White Cross Nursing Home, Higashimurayama, Tokyo, Japan